CLINICAL TRIAL: NCT05172414
Title: A Novel Fecal Sample Collection Method for Metagenomic Analyses
Status: Completed | Type: Observational
Sponsor: Onegevity Health (Industry)
Responsible Party: Sponsor
Other Study IDs: 002
Record Dates: First submitted 2021-12-02; First posted 2021-12-29 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: gut microbiome; metagenomic sequencing; stool collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Metagenomic (DNA) analysis of (stool) gut microbiome samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — The single group had no intervention. All followed the same procedures of different collection methods.

SUMMARY:
This is an open-label, one-arm, one-time-point pilot assessing the intra- and inter-group variation of gut microbiome collection methods and storage conditions using metagenomic sequencing for analysis. This study recruited 6 adult volunteers collecting 12 fecal samples from one bowel movement. Subjects were given detailed instructions as to collect and store feces samples into the 4 different collection and preservation methods and return samples for metagenomic analysis.

DETAILED DESCRIPTION:
A total of 6 subjects were enrolled in this pilot study. The inclusion criteria to be enrolled in the study included: age >18; Bristol Stool Scale type 3 and 4 (normal), agree to collect and donate the feces, and the ability to understand and write English. Exclusion criteria included people with constipation, slightly dry, or diarrhea feces (Bristol Stool Scale types 1-2, 5-7), pregnant or breastfeeding females, history of alcohol, drug, or medication abuse, known allergies to any substance in the study product, current diagnosis of inflammatory bowel disease (Crohn's Disease or Ulcerative Colitis), and currently taking any medication that may interfere with defecation.

Fecal collection kits were mailed to subjects with instructions for sample collection. A total of 12 samples (3 sites on the bowel movement, 4 collection/preserving methods) were collected by each subject yielding a total of 72 samples to be processed. Four preservation methods were used to process the samples for metagenomic sequencing: freezing (-20°C), room temperature storage, Zymo DNA shield kit (room temperature), and DESS DNA preservation (room temperature). All the samples are shipped at room temperature except the samples meant for freezing which were shipped on dry ice. At the lab, all the samples were put into a fridge (4°C) except the frozen samples which were put in a -20°C freezer.

Samples underwent DNA extraction and sequencing per previously published methods with the objective to understand intra- and inter-sample comparisons for collection methods and stability during storage/shipping. Results will include taxonomic abundance metrics, metabolic pathway classification, and diversity analysis.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adults, age ≥ 18 years 2. With normal to slightly diarrhea feces (Bristol Stool Scale - type 4 and type 5) 3. Agree to collect and donate the feces 4. Able to understand and write English 5. Voluntarily consent to the study and understand its nature and purpose including potential risks and side effects

Exclusion Criteria:

* 1. People with constipation, slightly dry or diarrhea feces (Bristol Stool Scale - type 1-3 and type 6-8) 2. Pregnant or breastfeeding females 3. History of alcohol, drug, or medication abuse 4. Known allergies to any substance in the study product 5. Current diagnosis of inflammatory bowel disease (Crohn's or Ulcerative Colitis) 6. Taking medication that may interfere with the defecation

Vulnerable Participants: No children, pregnant women, nursing home residents or other institutionalized persons, prisoners, or any other vulnerable participants were eligible to participate in this study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In order to account for potential drop-out, 6 participants were enrolled to achieve a properly-powered sample size. This target sample size was informed by the literature review and power analysis. Both males and females could participate, ages 18+, with no exclusions to race or ethnicity.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Dissolvable Wipe Comparison to Commercially Available Kits | 1 timepoint, 6 subjects, comparing the 4 collections in kits from a stool sample at 3 sites on a bowel movement. Each subject collected their sample on one day, and all samples were collected over one week.
  The primary outcome was is to assess the extent to which our novel approach to fecal sample collection (dissolvable wipe) and stabilization could maintain microbiota composition relative to immediate freezing (-20°C), preservation with a commercially available kit, and storage at room temperature (RT).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R. D'Adamo, PhD, Principal Investigator — University of Maryland
Locations (1):
- Center for Integrative Medicine at the University of Maryland School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- See also: Pre-print of this study (not peer-reviewed) — https://www.biorxiv.org/content/10.1101/2021.12.03.471072v1